CLINICAL TRIAL: NCT02157753
Title: Osteoporotic Fractures in a Swiss Trauma Center - Observational Study to Improve the Diagnosis and Management of and the Persistence to Therapy.
Brief Title: Quality of the Detection & Treatment of Osteoporotic Fractures in a Swiss Trauma Center
Status: Completed | Type: Observational
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Thomas Gross, MD, Prof. Dr. med., Kantonsspital Aarau
Other Study IDs: 2013/036
Record Dates: First submitted 2014-06-03; First posted 2014-06-06 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Osteoporosis, Postmenopausal; Osteoporosis
Keywords: Osteoporotic fracture; treatment for osteoporosis; adherence and compliance
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Osteoporotic Fractures; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
As a tertiary hospital the Traumatology department at the Kantonsspital Aarau looks after about 500 fracture patients hospitalized with an age over 50 years a year. First, we were interested in the effective rate of osteoporotic fractures in this cohort. As to this objective we offered subsequent diagnostics in suspected patients. 2012 we introduced a diagnostic pathway for every patient over 50 years of age with a fracture, including dual energy x-ray absorptiometry (DXA), a questionnaire about risk factors concerning osteoporosis and risk of fracture, the WHO Fracture Risk Assessment Tool (FRAX) and a laboratory workup focusing on this topic. Considering all these information we sent a detailed therapy-plan to the responsible General practitioner.

The main goal of this study is to verify the persistence and compliance of the osteoporosis therapy 12-15 months after fracture and to clarify any obstacles potentially impeding therapy (prejudice, adverse events, contraindication overlooked, financial problems etc.). The investigators use a postal questionnaire provided to the patient and the general practitioner. Data collection is undertaken by a study nurse, in addition phoning for missing data by phone-call. With the aim to ameliorate the implementation of treatment, patients and general practitioners will be provided with the specifically tailored information found to be missing.

ELIGIBILITY:
Inclusion criteria:

* age over 50 years
* any peripheral fracture, which led to hospitalisation in Kantonsspital Aarau, traumatology department

Exclusion Criteria:

* no informed consent
* age under 50 years
* not treated by traumatology department

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient with fracture over age of 49, admitted to the Kantonsspital Aarau and treated by the traumatology department, whom a treatment for osteoporosis was suggested according to national guidelines
Sampling Method: Non-Probability Sample
Enrollment: 478 (Actual)
Dates: Start 2012-07; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Persistence and compliance with treatment for osteoporosis | 12-15 month after initial fracture
  * percentage of persons receiving prescription vs. following completely / partially treatment advice
  * both, according to self declaration vs. general practitioner information
  * collection of arguments if therapy was not undertaken

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gross, Prof. Dr. med., Principal Investigator — Kantonsspital Aarau; Christoph Hemmeler, Dr.med., Principal Investigator — Kantonsspital Aarau
Locations (1):
- Kantonsspital Aarau, Aarau, Switzerland

REFERENCES:
- [Result] Morell S, Hemmeler C, Amsler F, Gross T. Adherence to osteoporosis pharmacotherapy one year after osteoporotic fracture - a Swiss trauma center secondary prevention project. Swiss Med Wkly. 2017 Jul 10;147:w14451. doi: 10.4414/smw.2017.14451. eCollection 2017. PMID 28695555
- [Result] Hemmeler C, Morell S, Amsler F, Gross T. Screening for osteoporosis following non-vertebral fractures in patients aged 50 and older independently of gender or level of trauma energy-a Swiss trauma center approach. Arch Osteoporos. 2017 Dec;12(1):38. doi: 10.1007/s11657-017-0334-3. Epub 2017 Apr 8. PMID 28391563